CLINICAL TRIAL: NCT04498702
Title: A Phase II Single-Arm, Open-Label, Multi-Center Study of Continuous APL-1202 Treatment in Subjects With High-Risk Non-Muscle-Invasive Bladder Cancer (NMIBC) Relapsed From Intravesical Chemo/BCG Therapy
Brief Title: Study of Continuous APL-1202 Treatment in Subjects With High-Risk Non-Muscle-Invasive Bladder Cancer (NMIBC) Relapsed From Intravesical Chemo/BCG Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Yahong Meditech Co., Ltd aka Asieris (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YHCT-1
Record Dates: First submitted 2020-07-22; First posted 2020-08-04 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-07

CONDITIONS: Non-muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APL-1202 treatment (Experimental)
  Interventions: Drug: APL-1202 treatment

INTERVENTIONS:
Drug: APL-1202 treatment — A modified 3+3 design was employed: The dose was started at 300 mg and increased to 450 mg, 600 mg and 750 mg if there was no dose-limiting toxicity (DLT) in 3 subjects after 4-week consecutive administration of APL-1202. When the dose-escalation study was in progress, the doses for any newly enrolled subjects would be the starting dose or the highest dose confirmed with no DLT by the dose-escalation cohort at the time of enrollment. When the MTD or the 750 mg daily dose was attained as a safe dose, the dose for all subjects in the study or subsequently enrolled subjects would be MTD or 750 mg/day.

SUMMARY:
To determine the efficacy of oral APL-1202 administered consecutively for 12 weeks in subjects with high-risk NMIBC relapsed from intravesical chemo/BCG therapy based on the recurrence-free rate (RFR) at 12 months after APL-1202 treatment.

DETAILED DESCRIPTION:
This trial was a single-arm, open-label, multi-center clinical study consisting of two periods: the dose-escalation and treatment period, and the follow-up and maintenance period.

Dose-Escalation and Treatment Period APL-1202 was orally administered TID daily and continuously for 12 weeks. APL-1202 dose was increased from daily 300, 450, 600 to 750mg or maximum tolerated dose (MTD).

A modified 3+3 design was employed: The dose was started at 300 mg and increased to 450 mg, 600 mg and 750 mg if there was no dose-limiting toxicity (DLT) in 3 subjects after 4-week consecutive administration of APL-1202. When the dose-escalation study was in progress, the doses for any newly enrolled subjects would be the starting dose or the highest dose confirmed with no DLT by the dose-escalation cohort at the time of enrollment. When the MTD or the 750 mg daily dose was attained as a safe dose, the dose for all subjects in the study or subsequently enrolled subjects would be MTD or 750 mg/day.

Follow-up and Maintenance Period APL-1202 was orally administered at the highest safe dose proven by the dose-escalation cohort, continuously for 3 months; This period was 12 months. To fit the 3-month cystoscopy follow-up schedule, the maintenance therapy, starting from 3-month off, was given continuously every other 3 months, resulting in 6 months of dosing in total.

APL-1202 daily administration schedule:

The first dose: within 30 minutes after breakfast; The second dose: within 30 minutes after lunch, and there should be a 4-hour interval between the first and second doses; The third dose: taken with a light snack at night before going to bed.

ELIGIBILITY:
Inclusion Criteria:

1. Well-informed with this trial and willing to sign the informed consent form;
2. Subjects have been clinically and histologically proven as relapsed high-risk non-muscle-invasive urothelial carcinoma of the bladder through clinical cystoscopy, urine cytology and pathological examination within 28 days before the enrollment; Subjects who met the high-risk definition in EAU Guidelines on Non-Muscle-Invasive Bladder Cancer (2012 Edition), including those who met the high-risk definition in current or any previous recurrence or primary diseases; Papillary carcinomas may or may not include Cis; All papillary carcinoma subjects with no visible tumor after transurethral resection of bladder tumor (TURBT); May include Cis subjects with visible tumors remaining after TURBT;
3. Past treatment history:

   Chemo-relapsed subgroup: the subjects who should have had intravesical chemotherapy in the 3 years prior to enrollment, but could not undergo any BCG therapy; BCG-relapsed subgroup: the subjects who should have had intravesical BCG treatment in the 3 years prior to enrollment, prior intravesical chemotherapy is allowed;
4. Subjects with treatment failure included:

   Subjects with recurrence after at least one intravesical course; BCG-relapsed subjects might include those intolerable to intravesical BCG therapy; Subjects with tumor grade progression after intravesical therapy;
5. The subject is willing to provide cystoscopic biopsy specimens for assessment
6. Age ≥ 18 years, male or female;
7. Performance status score (ECOG scale) ≤ 1 (0-1), and did not deteriorate within 7 days;
8. The subject must have normal organ and bone marrow functions within 28 days prior to enrollment into the study (based on normal range measured by the clinical site):

   ANC > 1.0×109 /L; Platelet count > 100×109 /L; Hemoglobin > 9.0 g/dL; ALP < 2.5 times upper limit of normal range (should be less than 10 times upper limit of normal range if at the presence of bone metastasis); GFR (calculated using Cockcroft-Gault formula) ≥ 50 mL/min; INR < 1.5, except subjects who was undergoing Warfarin treatment at the time of screening.
9. Subjects who were receiving other medications with known or potential effects on the efficacy or pharmacokinetics of nitroxoline should be assessed and determined by the principal investigator.
10. Female subjects must be surgically sterilized or menopaused or must agree to take effective contraceptive measures during the treatment. Male subjects must be surgically sterilized or must agree to take effective contraceptive measures during treatment. Subjects must continue to take contraceptive measures for 3 months after the investigational therapy was completed. Definition of an effective contraceptive measure should be determined at the discretion of the principal investigator or any investigator appointed by the principal investigator.
11. Life expectancy is over 12 months.

Exclusion Criteria:

1. TBIL, ALT or AST exceeded 1.5 times upper limit of the normal range (based on the normal range determined by the clinical site);
2. Upper tract urothelial carcinoma;
3. Subjects who had systemic chemotherapy on bladder carcinoma in the past;
4. Subject who had undergone any surgical procedure (excluding TURBT or cystoscopy), radiotherapy or systemic chemotherapy within 4 weeks prior to enrollment;
5. Grade 3 hemorrhage as per NCI CTCAE 4.0 occurred within 4 weeks prior to enrollment;
6. Any of the following conditions occurred within 6 months prior to enrollment: myocardial infarction, serious/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism;
7. Regardless of antihypertensive medication, systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg;
8. Subjects having a malignancy history within 2 years, except cured basal cell carcinoma, squamous cell skin cancer or cervical carcinoma "in situ";
9. Subjects with any optic nerve disorder or having a history of optic nerve disorders;
10. Subjects with clinically uncontrolled active infections such as acute pneumonia, immunoactive phase of hepatitis B, etc.;
11. Subjects with dysphagia or any known drug absorption disorder;
12. Subjects with anuria;
13. Subjects with any active digestive disease such as duodenal ulcer and ulcerative colitis or any other conditions potentially leading to gastrointestinal hemorrhage or perforation as identified by the investigator;
14. The investigator deemed that a subject might have increased risk for the study or medication or had any other serious acute or chronic medical conditions potentially interfering with interpretation and judgment of study results;
15. Any pregnant or breastfeeding woman or any woman with a positive pregnancy test results prior to the first medication;
16. Subjects having a serious mental disorder with compliance concern in this clinical study;
17. Subjects participating in any other clinical drug trial in the past 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-05-13 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-01-18 (Actual)

PRIMARY OUTCOMES:
Recurrence-free rate (RFR) at the end of 12-month follow-up in subjects with high-risk NMIBC relapsed from intravesical chemo/BCG therapy. | 12 months
  Recurrence-free rate (RFR) at the end of 12-month follow-up in subjects with high-risk NMIBC relapsed from intravesical chemo/BCG therapy.

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | 12 months
  Recurrence-free survival (RFS)
Progression-free survival (PFS). | 12 months
  progression-free survival (PFS).
The safety and tolerability of APL-1202. | 12 months
  Post-medication safety assessment included laboratory parameters, physical examination, vital signs, performance status score, and AEs. Frequency and severity of AEs were rated in accordance with internationally agreed NCI CTC AE4.0.
Plasma Max Concentration - APL-1202 and its metabolites | Day 28
  PK measurement expressed as maximum plasma concentration for APL-1202 and metabolites
Plasma Steady state Concentration - APL-1202 and its metabolites | Day 28
  PK measurement expressed as Steady state Concentration for plasma APL-1202 and its metabolites
Plasma Area Under Curve - APL-1202 and its metabolites | Day 28
  PK measurement expressed as area under curve for plasma APL-1202 and its metabolites
Urinary excreted amounts- APL-1202 and its metabolites | Day 28
  PK measurement expressed as Urinary excreted amounts for APL-1202 and its metabolites
Cumulative urinary excreted amounts- APL-1202 and its metabolites | Day 28
  PK measurement expressed as Cumulative Urinary excreted amounts for APL-1202 and its metabolites
Cumulative fraction of dose- APL-1202 and its metabolites | Day 28
  PK measurement expressed as Cumulative fraction of dose for APL-1202 and its metabolites
The SNV(single-nucleotide variant) patterns of bladder cancer related genes in pre- and post-treatment plasma ctDNA (circulating tumor DNA) through targeted amplicon sequencing | 12 months
  Blood ctDNA were extracted from the patients before APL-1202 treatment or after APL-1202 treatment; somatic SNV were detected by targeted amplicon sequencing. Evaluation of RFR (Recurrence-free rate), RFS (Recurrence-free survival), PFS (Progression-free survival) and baseline SNV will be performed using cox regression survival model.
The InDel (insertion-deletion) patterns of bladder cancer related genes in pre- and post-treatment plasma ctDNA (circulating tumor DNA) through targeted amplicon sequencing | 12 months
  Blood ctDNA were extracted from the patients before APL-1202 treatment or after APL-1202 treatment; somatic InDel were detected by targeted amplicon sequencing. Evaluation of RFR (Recurrence-free rate), RFS (Recurrence-free survival), PFS (Progression-free survival) and baseline InDel will be performed using cox regression survival model.

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, MD,PhD, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No